CLINICAL TRIAL: NCT00355173
Title: Pilot Study to Assess the Efficacy and Safety of the Lubo Cervical Collar
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Arik Tzukert, DMD
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB001-HMO-CTIL
Record Dates: First submitted 2006-07-20; First posted 2006-07-21 (Estimated); Last update posted 2011-05-12 (Estimated); Status verified 2010-02

CONDITIONS: Elective Surgical Procedure

INTERVENTIONS:
Device: Lubo cervical collar

SUMMARY:
The Lubo cervical collar is a device that simultaneously maintains cervical spine control and keeps an open airway in a non-invasive manner. The purpose of the device is to manage cervical spine control and airway protection in the trauma patient.

DETAILED DESCRIPTION:
Cervical spine stabilization is usually achieved by a semi-rigid collar. While these collars achieve the goal of supporting the cervical spine, they limit the possibilities for jaw thrust or other airway manipulations. Definitive airway protection usually must be achieved by orotracheal intubation. Thee Lubo collar is a device that simultaneously maintains cervical spine control and keeps an open airway in a non-invasive manner that is simple to operate. The objective of the study is to test the safety of the collar volunteers. The study is composed of two stages:1.healthy volunteers that will not undergo any intervention except testing the LCC.2. second group of patients scheduled to undergo an operation under general anesthesia with endotracheal intubation or laryngeal mask airway.

ELIGIBILITY:
Inclusion criteria

1. Males or females.
2. Age 18-60.
3. Normal airway anatomy, with expected easy ventilation and intubation.
4. Anesthetic risk- class 1or 2 by the American Society of Anesthesiologists (ASA) criteria.
5. Patients scheduled for an elective operation at the lower part of the body in supine position not supposed to last more then 2 hours.
6. Anesthetic plan- general anesthesia

Exclusion criteria

1. Known problems of the cervical spine.
2. Known problems of the temporomandibular joint.
3. Suspected difficult intubation or difficult mask ventilation.
4. High risk of gastric content aspiration.
5. Morbid obesity (BMI >32).
6. Pregnancy
7. Psycho- social problems
8. Any cerebrovascular or cardiovascular disease
9. Known hypersensitivity reactions to fabrics or plastics
10. Any rash, eruption, wounds or sores at the upper torso, the neck and the head.
11. No participation in other clinical trail at the time of the trail

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-05; Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Omri Lubovsky, M.D., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Lubovsky O, Liebergall M, Weissman C, Yuval M. A new external upper airway opening device combined with a cervical collar. Resuscitation. 2010 Jul;81(7):817-21. doi: 10.1016/j.resuscitation.2010.02.013. Epub 2010 Apr 20. PMID 20409626